CLINICAL TRIAL: NCT04888585
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of ABBV-154 in Subjects With Moderately to Severely Active Rheumatoid Arthritis With Inadequate Response to Biologic and/or Targeted Synthetic Disease-Modifying Anti-Rheumatic Drugs (b/tsDMARDs)
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity in Participants Between 18 to 75 Years of Age Treated With Subcutaneous (SC) Injections of ABBV-154 for Moderately to Severely Active Rheumatoid Arthritis (RA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M20-466; 2020-005303-39 (EudraCT Number)
Record Dates: First submitted 2021-05-13; First posted 2021-05-17 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); ABBV-154; AIM-RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose A of ABBV-154 (Experimental): Participants in this group will receive dose A of ABBV-154 subcutaneously (SC) every other week (eow) for 12 weeks in the placebo-controlled period, 66 weeks in the long term extension (LTE) period 1 and 104 weeks in LTE period 2.
  Interventions: Drug: ABBV-154
- Dose B of ABBV-154 (Experimental): Participants in this group will receive dose B of ABBV-154 SC eow for 12 weeks in the placebo-controlled period, 66 weeks in the LTE period 1 and 104 weeks in LTE period 2.
  Interventions: Drug: ABBV-154
- Dose C of ABBV-154 EOW (Experimental): Participants in this group will receive dose C of ABBV-154 SC eow for 12 weeks in the placebo-controlled period, 66 weeks in the LTE period 1 and 104 weeks in LTE period 2.
  Interventions: Drug: ABBV-154
- Dose C of ABBV-154 E4W (Experimental): Participants in this group will receive dose C of ABBV-154 SC every 4 weeks (e4w) for 12 weeks in the placebo-controlled period, 66 weeks in the LTE period 1 and 104 weeks in LTE period 2.
  Interventions: Drug: ABBV-154
- Placebo (Experimental): Participants in this group will receive placebo SC eow for 12 weeks in the placebo-controlled period and will be re-randomized in 1:1 ratio to receive ABBV-154 dose B or C respectively SC eow for 66 weeks in the LTE period 1 and 104 weeks in LTE period 2.
  Interventions: Drug: ABBV-154; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-154 — Subcutaneous Injection
Drug: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
Rheumatoid Arthritis (RA) is an inflammatory disease of the joints causing pain, stiffness, swelling and loss of joint function. This study evaluated how safe and effective ABBV-154 is in participants treated for moderately to severely active RA. Adverse events and change in the disease activity were assessed.

ABBV-154 is an investigational drug being evaluated for the treatment of RA. Study doctors placed the participants in 1 of 5 treatment groups or arms; each arm received a different treatment. There was a 1 in 5 chance that participants were assigned to placebo. Participants 18-75 years of age with moderate to severe RA were enrolled. Around 425 participants were to be enrolled in the study at approximately 270 sites worldwide.

The study was comprised of a 12 week placebo-controlled period, a double-blind long term extension (LTE) period 1 of 66 weeks, a LTE period 2 of 104 weeks and a follow-up visit 70 days after the last dose of the study drug. In the LTE period 1, participants in the placebo group were re-randomized to receive ABBV-154 at 1 of 2 different doses SC every other week (EOW). Other participants remained on their previous dose and dosing regimen of ABBV-154.

There may have been a higher treatment burden for participants in this trial compared to their standard of care. Participants attended regular visits during the study at a hospital or clinic. The effect of the treatment was checked by medical assessments, blood tests, and side effects, and completing questionnaires.

DETAILED DESCRIPTION:
Participants were randomly assigned at a ratio of 1:1:1:1:1 to ABBV-154 at either 40 mg, 150 mg, 340 mg, subcutaneously (SC) EOW; 340 mg SC every 4 weeks (E4W); or placebo SC EOW. Randomization was stratified by baseline glucocorticoid (yes/no); number of prior failed biologic and/or targeted synthetic disease-modifying anti-rheumatic drugs (b/tsDMARDs) (1; 2 or more); and prior anti-TNF failure (yes/no) and if yes, further stratification by prior adalimumab use (yes/no).

After 12 weeks, participants receiving placebo were re-randomized to receive ABBV-154 150 mg SC EOW or 340 mg SC EOW for the long-term extension (LTE) periods. At re-randomization, participants were stratified by baseline glucocorticoid use (yes/no) and prior adalimumab use (yes/no). Participants from the other dose groups were to continue with their respective dose and dosing regimen.

The primary analysis was conducted after all ongoing participants completed Week 12 or withdrew from the study. A final analysis was to be conducted after all participants completed LTE period 2 and a safety follow-up visit or withdrew from the study. The study was terminated before any participants entered LTE Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis(RA) with fulfillment of the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA.
* Participant has >= 6 swollen joints (based on 66 joint count) and >=6 tender joints (based on 68 joint count) at baseline.
* Participant must have had an inadequate response to at least one prior biologic and/or targeted synthetic disease-modifying anti-rheumatic drugs (b/tsDMARDs) treatment for RA.
* Participants must be on stable dose of methotrexate (MTX).

Exclusion Criteria:

- Participant discontinued prior adalimumab therapy due to intolerability or toxicity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (220):
- United States (101):
  - Elite Clinical Studies, LLC /ID# 228227, Phoenix, Arizona
  - Arthritis and Rheumatism Associates /ID# 228201, Jonesboro, Arkansas
  - Providence Medical Foundation /ID# 228104, Fullerton, California
  - Care Access Research, Huntington Beach /ID# 228163, Huntington Beach, California
  - Purushotham & Akther Kotha MD, Inc /ID# 228120, La Mesa, California
  - Arthritis & Osteo Medical Ctr /ID# 228239, La Palma, California
  - Pacific Arthritis Care Center - Los Angeles /ID# 229330, Los Angeles, California
  - California Medical Research Associates /ID# 230131, Northridge, California
  - Arthritis Care And Research Center ACRC /ID# 230099, Poway, California
  - East Bay Rheumatology Medical /ID# 228099, San Leandro, California
  - Millennium Clinical Trials /ID# 230618, Thousand Oaks, California
  - The Lundquist Institute at Harbor-UCLA Medical Center /ID# 228241, Torrance, California
  - Medvin Clinical Research /ID# 228181, Tujunga, California
  - Inland Rheum & Osteo Med Grp /ID# 228204, Upland, California
  - Comprehensive Rheumatology Center /ID# 230132, Woodland Hills, California
  - Denver Arthritis Clinic /ID# 228172, Denver, Colorado
  - New England Research Associates, LLC /ID# 230127, Bridgeport, Connecticut
  - Stamford Therapeutics Consorti /ID# 229214, Stamford, Connecticut
  - Delaware Arthritis /ID# 229413, Lewes, Delaware
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 228229, Boca Raton, Florida
  - Bay Area Arthritis and Osteo /ID# 228075, Brandon, Florida
  - Clinical Research of West Florida, Inc /ID# 228128, Clearwater, Florida
  - International Medical Research /ID# 228069, Daytona Beach, Florida
  - Omega Research Debary, LLC /ID# 228293, DeBary, Florida
  - Neoclinical Research /ID# 228753, Hialeah, Florida
  - University of Florida /ID# 228242, Jacksonville, Florida
  - Lakes Research, LLC /ID# 228665, Miami, Florida
  - University of Miami /ID# 228737, Miami, Florida
  - Suncoast Clinical Research /ID# 228237, New Port Richey, Florida
  - Omega Research Group /ID# 229966, Orlando, Florida
  - HMD Research LLC /ID# 228185, Orlando, Florida
  - Millennium Research /ID# 228183, Ormond Beach, Florida
  - Arthritis Center, Inc. /ID# 228209, Palm Harbor, Florida
  - BayCare Medical Group /ID# 228289, St. Petersburg, Florida
  - West Broward Rheumatology Associates /ID# 228603, Tamarac, Florida
  - Clinical Research of West Florida - Tampa /ID# 228186, Tampa, Florida
  - Conquest Research /ID# 230560, Winter Park, Florida
  - Florida Medical Clinic /ID# 228236, Zephyrhills, Florida
  - Arthritis and Rheumatology /ID# 228743, Atlanta, Georgia
  - Jefrey D. Lieberman, MD, P.C. /ID# 230129, Decatur, Georgia
  - Arthritis Center of North GA /ID# 228769, Gainesville, Georgia
  - Atlanta Research Center for Rheumatology /ID# 230430, Marietta, Georgia
  - Great Lakes Clinical Trials /ID# 228699, Chicago, Illinois
  - Greater Chicago Specialty Physicians /ID# 228282, Schaumburg, Illinois
  - Clinic of Robert Hozman/Clinical Investigation Specialists /ID# 228174, Skokie, Illinois
  - Springfield Clinic /ID# 228124, Springfield, Illinois
  - Beacon Medical Group Clinical Research /ID# 229153, Granger, Indiana
  - University of Iowa Hospitals and Clinics /ID# 229217, Iowa City, Iowa
  - Four Rivers Clinical Research /ID# 230109, Paducah, Kentucky
  - The Arthritis & Diabetes Clinic, Inc. /ID# 228221, Monroe, Louisiana
  - Klein and Associates MD /ID# 230145, Cumberland, Maryland
  - Klein and Associates MD - Hagerstown /ID# 230143, Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research /ID# 228617, Wheaton, Maryland
  - AA Medical Research Center - Grand Blanc /ID# 228604, Grand Blanc, Michigan
  - Advanced Rheumatology, PC /ID# 228684, Lansing, Michigan
  - June DO, PC /ID# 229838, Lansing, Michigan
  - Arthritis Associates /ID# 230188, Hattiesburg, Mississippi
  - Rheumatology Consultants - Clinical Research /ID# 229208, Tupelo, Mississippi
  - Clayton Medical Associates, P.C. dba Saint Louis Rheumatology /ID# 228283, St Louis, Missouri
  - West County Rheumatology /ID# 228102, St Louis, Missouri
  - Logan Health Research /ID# 228273, Kalispell, Montana
  - Advanced Biomedical Research of America /ID# 228596, Las Vegas, Nevada
  - Innovative Health Research /ID# 229209, Las Vegas, Nevada
  - Arthritis and Osteoporosis Associates /ID# 229418, Freehold, New Jersey
  - Arthritis Rheumatic and Back Disease Associates. P.A. /ID# 228602, Voorhees Township, New Jersey
  - Albuquerque Center For Rheumatology /ID# 228709, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Inc /ID# 228925, Albuquerque, New Mexico
  - Arthritis and Osteo Assoc /ID# 228662, Las Cruces, New Mexico
  - Buffalo Rheumatology and Medicine - Orchard Park /ID# 228710, Orchard Park, New York
  - St. Lawrence Health System /ID# 229508, Potsdam, New York
  - DJL Clinical Research, PLLC /ID# 230133, Charlotte, North Carolina
  - Cape Fear Arthritis Care /ID# 228747, Leland, North Carolina
  - PMG Research of Salisbury /ID# 230627, Salisbury, North Carolina
  - Trinity Health Med Arts Clinic /ID# 228202, Minot, North Dakota
  - University of Cincinnati /ID# 229212, Cincinnati, Ohio
  - Paramount Medical Research Con /ID# 228254, Middleburg Heights, Ohio
  - Arthritis Assoc of NW Ohio /ID# 228936, Toledo, Ohio
  - Arthritis and Rheumatology Center of Oklahoma /ID# 228975, Oklahoma City, Oklahoma
  - Rheumatology Associates of Oklahoma /ID# 228701, Oklahoma City, Oklahoma
  - Advanced Rheumatology & Arthritis Wellness Center /ID# 228608, Cranberry Township, Pennsylvania
  - Altoona Ctr Clinical Res /ID# 230058, Duncansville, Pennsylvania
  - Arthritis Group /ID# 229777, Philadelphia, Pennsylvania
  - PA Regional Center for Arthritis and Osteoporosis Research /ID# 228742, Wyomissing, Pennsylvania
  - Columbia Arthritis Center /ID# 228705, Columbia, South Carolina
  - West Tennessee Research Institute /ID# 228257, Jackson, Tennessee
  - Arthritis and Rheumatology Research Institute, PLLC /ID# 228937, Allen, Texas
  - Allen Arthritis /ID# 228712, Allen, Texas
  - Trinity Universal Research Associates - Carrollton /ID# 230104, Carrollton, Texas
  - Adriana Pop-Moody MD Clinic PA /ID# 230062, Corpus Christi, Texas
  - West Texas Clinical Research /ID# 228276, Lubbock, Texas
  - P&I Clinical Research /ID# 230183, Lufkin, Texas
  - SW Rheumatology Res. LLC /ID# 228088, Mesquite, Texas
  - Trinity Universal Research Associates, Inc /ID# 228238, Plano, Texas
  - Epic Medical Research /ID# 228097, Red Oak, Texas
  - Sun Research Institute /ID# 228768, San Antonio, Texas
  - Advanced Rheumatology of Houston /ID# 228170, The Woodlands, Texas
  - DM Clinical Research - Tomball /ID# 228112, Tomball, Texas
  - Rheumatology Clinic of Houston /ID# 228178, Tomball, Texas
  - Arthritis & Osteoporosis Clinic /ID# 228736, Waco, Texas
  - Tidewater Physicians Medical Center /ID# 230130, Newport News, Virginia
  - Arthritis Northwest, PLLC /ID# 228275, Spokane, Washington
- Australia (5):
  - Emeritus Research Sydney /ID# 230070, Botany, New South Wales
  - BJC Health /ID# 229015, Paramatta, New South Wales
  - Rheumatology Research Unit Sunshine Coast /ID# 229017, Maroochydore, Queensland
  - The Queen Elizabeth Hospital /ID# 230071, Woodville South, South Australia
  - Emeritus Research /ID# 229018, Camberwell, Victoria
- Canada (5):
  - Rheumatology Research Associates /ID# 227818, Edmonton, Alberta
  - Manitoba Clinic /ID# 227822, Winnipeg, Manitoba
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 227821, Sainte-Foy, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 227824, Trois-Rivières, Quebec
  - Dr Naik-Medical Professional Corporation-Alliance Health /ID# 227823, Saskatoon, Saskatchewan
- Czechia (6):
  - Revmatologicky ustav v Praze /ID# 229188, Prague
  - PV MEDICAL Services s.r.o. /ID# 228265, Prague
  - Revmatologicka ambulance - MUDr. Zuzana Urbanova /ID# 227775, Prague
  - Fakultni Nemocnice v Motole /ID# 231622, Prague
  - MEDICAL PLUS, s.r.o. /ID# 228030, Uherské Hradiště
  - RHEUMA s.r.o. /ID# 230850, Velké Bílovice
- Germany (3):
  - Rheumazentrum Ruhrgebiet /ID# 227850, Herne, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 229526, Berlin
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH /ID# 227785, Hamburg
- Greece (4):
  - General Hospital of Athens Gennimatas /ID# 227806, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 227804, Heraklion, Crete
  - 424 General MILITARY Hospital /ID# 227805, Efkarpia (Thessalonikis), Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 229614, Thessaloniki
- Hungary (8):
  - Debreceni Egyetem Klinikai Kozpont /ID# 228371, Debrecen, Hajdú-Bihar
  - Obudai Egeszsegugyi Centrum Kft. /ID# 228359, Budapest, Pest County
  - DRC Gyogyszervizsgalo Kozpont Kft /ID# 228365, Balatonfüred
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 227671, Budapest
  - Revita Reumatologiai Rendelo /ID# 227668, Budapest
  - CMED Rehabilitacios es Diagnosztikai Kozpont /ID# 227670, Székesfehérvár
  - Vital Medical Center Orvosi es Fogaszati Kozpont (Vital Medicina Kft.) /ID# 227669, Veszprém
  - Obudai Egeszsegugyi Centrum Kft. Zalaegerszeg /ID# 228374, Zalaegerszeg
- Israel (6):
  - Meir Medical Center /ID# 226800, Kfar Saba, Central District
  - Rambam Health Care Campus /ID# 226798, Haifa, H_efa
  - Bnai Zion Medical Center /ID# 226801, Haifa, H_efa
  - The Lady Davis Carmel Medical Center /ID# 226802, Haifa, H_efa
  - The Chaim Sheba Medical Center /ID# 226797, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 228341, Tel Aviv, Tel Aviv
- Italy (3):
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma /ID# 228917, Rome, Lazio
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 228581, Ancona
  - Azienda Ospedaliera Universitaria Paolo Giaccone /ID# 228583, Palermo
- Japan (23):
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital /ID# 229899, Nagoya, Aichi-ken
  - Daido Clinic /ID# 229280, Nagoya, Aichi-ken
  - Sugimoto rheumatology and internal medicine clinic /ID# 229495, Fukui-shi, Fukui
  - Hamanomachi Hospital /ID# 228644, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center /ID# 228642, Fukuoka, Fukuoka
  - Shono Rheumatism Clinic /ID# 229054, Fukuoka, Fukuoka
  - Katayama Orthopedic Rheumatology Clinic /ID# 229277, Asahikawa-shi, Hokkaido
  - Sagawa Akira Rheumatology Clin /ID# 228787, Sapporo, Hokkaido
  - Matsubara Mayflower Hospital /ID# 228948, Kato-shi, Hyōgo
  - Sanuki Municipal Hospital /ID# 229276, Sanuki-shi, Kagawa-ken
  - Bay Side Misato Medical Center /ID# 228947, Kochi, Kochi
  - Kumamoto Orthopaedic Hospital /ID# 228641, Kumamoto, Kumamoto
  - Medical Corporation Keiai Kai Clinic /ID# 228547, Miyazaki, Miyazaki
  - Sasebo Chuo Hospital /ID# 229168, Sasebo-shi, Nagasaki
  - Nagaoka Red Cross Hospital /ID# 229962, Nagaoka-shi, Niigata
  - National Hospital Organization Osaka Minami Medical Center /ID# 229174, Kawachinagano Shi, Osaka
  - Osaka City General Hospital /ID# 228786, Osaka, Osaka
  - Japanese Red Cross Osaka Hospital /ID# 229816, Osaka, Osaka
  - Azuma Rheumatology Clinic /ID# 230078, Sayama-shi, Saitama
  - St.Luke's International Hospital /ID# 229492, Chuo-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center /ID# 228720, Meguro-ku, Tokyo
  - Medical Corporation Uchida Clinic /ID# 229494, Sumida-ku, Tokyo
  - Tokito Clinic Rheumatology and Orthopaedics Surgery /ID# 228354, Shimonoseki-shi, Yamaguchi
- Netherlands (2):
  - Academisch Medisch Centrum /ID# 227234, Amsterdam
  - Maastricht Universitair Medisch Centrum /ID# 227235, Maastricht
- New Zealand (3):
  - Aotearoa Clinical Trials /ID# 229012, Papatoetoe, Auckland
  - Timaru Medical Specialists Ltd /ID# 229013, Timaru, Canterbury
  - Wellington Regional Hospital /ID# 233517, Newtown, Wellington Region
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela /ID# 227939, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 227170, Warsaw, Masovian Voivodeship
  - SANUS Szpital Specjalistyczny /ID# 227171, Stalowa Wola, Podkarpackie Voivodeship
  - ClinicMed Daniluk, Nowak Sp.k. /ID# 227919, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 228047, Gdansk, Pomeranian Voivodeship
  - MICS Centrum Medyczne Warszawa /ID# 231133, Warsaw
  - AMICARE Sp. z o.o. sp.k. /ID# 231327, Lodz, Łódź Voivodeship
- Puerto Rico (2):
  - GCM Medical Group PSC /ID# 228981, San Juan
  - Mindful Medical Research /ID# 228982, San Juan
- Russia (7):
  - LLC Family Outpatient Clinic No /ID# 227926, Korolev, Moscow
  - Moscow Regional Research and Clinical Institute n.a. Vladimirskiy (MONIKI) /ID# 228755, Moscow, Moscow Oblast
  - Family Clinic /ID# 227929, Yekaterinburg, Sverdlovsk Oblast
  - Kazan State Medical University /ID# 227927, Kazan', Tatarstan, Respublika
  - Central Clinical Hospital of Russian Academy of Science /ID# 229438, Moscow
  - Euromedservice /ID# 227933, Pushkin
  - Clinical Rheumatologic Hospital No 25 /ID# 227922, Saint Petersburg
- Slovakia (5):
  - MEDMAN s.r.o. /ID# 227826, Martin
  - Reum.hapi s.r.o. /ID# 227825, Nové Mesto nad Váhom
  - Thermium s.r.o. /ID# 227816, Piešťany
  - REUMAMED POPRAD s.r.o. /ID# 229628, Poprad
  - Reumex, s.r.o. /ID# 227827, Rimavská Sobota
- South Korea (6):
  - SoonChunHyang University CheonAn Hospital /ID# 228146, Cheonan-si, Chungcheongnam-do
  - Yonsei University Health System Severance Hospital /ID# 227659, Seoul, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospital /ID# 227658, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Hospital /ID# 227657, Daegu
  - Inha University Hospital /ID# 227656, Incheon
  - Asan Medical Center /ID# 227655, Seoul
- Spain (9):
  - Hospital Clínico Universitario de Santiago-CHUS /ID# 227420, Santiago de Compostela, A Coruna
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 227666, Sabadell, Barcelona
  - Hospital Universitario Basurto /ID# 227667, Bilbao, Vizcaya
  - Hospital Universitario A Coruna - CHUAC /ID# 227419, A Coruña
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 234115, Madrid
  - Hospital Universitario 12 de Octubre /ID# 227743, Madrid
  - Hospital Regional Universitario de Malaga /ID# 227418, Málaga
  - Hospital Universitario Virgen de Valme /ID# 227417, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 227408, Valencia
- Taiwan (4):
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation /ID# 227220, Chiayi City
  - Far Eastern Memorial Hospital /ID# 227373, New Taipei City
  - National Taiwan University Hospital /ID# 230001, Taipei
  - Taipei Veterans General Hosp /ID# 227376, Taipei
- Turkey (Türkiye) (3):
  - Hacettepe Universitesi Tip Fak /ID# 227796, Sihhiye, Ankara
  - Ankara Univ Medical Faculty /ID# 227797, Ankara
  - Kocaeli University Med Faculty /ID# 228244, Kocaeli
- Ukraine (8):
  - MNI City Multidisciplinary Hospital #18 Kharkiv City Council /ID# 228961, Kharkiv
  - Khmelnytskyi Regional Hospital /ID# 230680, Khmelnytskyi
  - Medical Center of Medical Clinic Blagomed LLC /ID# 228956, Kyiv
  - Medical Center "OK! Clinic+" LLC, "International Institute of Clinical Research" /ID# 228958, Kyiv
  - Medical Center CONSILIUM MEDICAL /ID# 228959, Kyiv
  - PI "Poltava Regional Clinical Hospital n.a. M.V.Sklifosovsky of PCC" /ID# 228962, Poltava
  - CNE Vinnytsya Regional Clinical Hospital named after N.I.Pirogov /ID# 228954, Vinnytsia
  - Сlinic Scientific Research Inst of Invalid Rehab ESMС M I Pyrogov VNMU /ID# 228955, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 473 participants (All Randomized Population) were enrolled in the study.
Pre-assignment Details: The ITT Population included all participants who were randomized and received at least 1 dose of study drug. One randomized participant (ABBV-154 150 mg EOW) was not treated and thus not included in the ITT population (N=472).
Groups:
- Period 1 (Placebo-Controlled Period) Placebo: Participants in this group received placebo subcutaneously (SC) every other week (EOW) for 12 weeks in the placebo-controlled period and were re-randomized at 1:1 ratio to receive ABBV-154 150 mg or 340 mg SC EOW for 66 weeks in the long term extension (LTE) period.
- Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Period 2 (Extension Period) ABBV-154 40 mg EOW: Participants in this group received 40 mg of ABBV-154 SC EOW for 12 weeks in the placebo-controlled period and 66 weeks in the LTE period.
- Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Period 2 (Extension Period) ABBV-154 150 mg EOW: Participants in this group received 150 mg of ABBV-154 SC EOW for 12 weeks in the placebo-controlled period and 66 weeks in the LTE period.
- Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Period 2 (Extension Period) ABBV-154 340 mg EOW: Participants in this group received 340 mg of ABBV-154 SC EOW for 12 weeks in the placebo-controlled period and 66 weeks in the LTE period.
- Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W: Participants in this group received 340 mg of ABBV-154 SC every 4 weeks (E4W) for 12 weeks in the placebo-controlled period and 66 weeks in the LTE period.
- Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW: Participants in this group received placebo SC EOW for 12 weeks in the placebo-controlled period and were re-randomized at 1:1 ratio to receive ABBV-154 150 mg or 340 mg SC EOW for 66 weeks in the LTE period.
- Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW: Participants in this group received placebo SC eow for 12 weeks in the placebo-controlled period and were re-randomized in 1:1 ratio to receive ABBV-154 150 mg or 340 mg respectively SC EOW for 66 weeks in the LTE period.
- Period 2 (Extension Period) ABBV-154 340 mg E4W: Participants in this group received 340 mg of ABBV-154 SC E4W for 12 weeks in the placebo-controlled period and 66 weeks in the LTE period.
Period: Placebo-Controlled (Baseline-Week 12)
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W | Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW | Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW | Period 2 (Extension Period) ABBV-154 40 mg EOW | Period 2 (Extension Period) ABBV-154 150 mg EOW | Period 2 (Extension Period) ABBV-154 340 mg EOW | Period 2 (Extension Period) ABBV-154 340 mg E4W
Started | 96 | 98 | 95 (One randomized participant was ineligible and did not receive treatment. This participant was was not included in the ITT population.) | 90 | 94 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 92 | 93 | 86 | 85 | 89 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 9 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 4 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long Term Extension (Wk 13-End of Study)
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W | Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW | Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW | Period 2 (Extension Period) ABBV-154 40 mg EOW | Period 2 (Extension Period) ABBV-154 150 mg EOW | Period 2 (Extension Period) ABBV-154 340 mg EOW | Period 2 (Extension Period) ABBV-154 340 mg E4W
Started | 0 | 0 | 0 | 0 | 0 | 45 (One participant from Period 1 Placebo group did not enter Period 2.) | 46 | 93 | 86 | 85 | 89
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 45 | 46 | 93 | 86 | 85 | 89
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 8 | 8 | 8 | 11
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 37 | 36 | 78 | 71 | 71 | 72
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 5 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) Population included all participants who were randomized and received at least 1 dose of study drug (N=472). The ITT Population was used for all efficacy analyses.
  The Placebo group from Period 1 was re-randomized to either 150 mg or 340 mg for the Long-Term Extension Periods 1 and 2. For the other groups from Period 1 receiving ABBV-154, participants continued receiving ABBV-154 at the same dose and dosing regimen as in Period 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W | Total
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94 | 472
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (11.28) | 56.2 (10.17) | 56.8 (9.91) | 59.5 (10.72) | 57.9 (10.70) | 57.6 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 73 | 70 | 74 | 373
  Male | 16 | 22 | 21 | 20 | 20 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 12 | 18 | 17 | 82
  Not Hispanic or Latino | 79 | 80 | 82 | 72 | 77 | 390
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 14 | 15 | 12 | 20 | 14 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 10 | 4 | 6 | 3 | 2 | 25
  White | 72 | 79 | 75 | 67 | 76 | 369
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Achievement of 50% Improvement as Measured by American College of Rheumatology Response Criteria (ACR50) at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician's Global Assessment of Disease Activity (NRS)
     * Patient's Global Assessment of Disease Activity (NRS)
     * Patient's Assessment of Pain (NRS)
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Week 12
Population: ITT analysis set participants were included (N=472); Participants with missing Week 12 data for reasons other than COVID-19 or logistical restrictions were counted as non-responders (non-responder imputation), unless they were a responder before and after Week 12 (responder imputation); participants with missing Week 12 data because of COVID-19 or logistical restrictions were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
Percentage of participants | 6.3 [1.4 to 11.1] | 25.5 [16.9 to 34.1] | 33.3 [23.7 to 42.9] | 44.4 [34.2 to 54.7] | 30.9 [21.5 to 40.2]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 21.2, 95% CI 2-sided [11.5 to 31.0] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 26.6, 95% CI 2-sided [16.5 to 36.7] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 37.7, 95% CI 2-sided [27.4 to 48.1] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 23.2, 95% CI 2-sided [13.8 to 32.6] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

2. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28 (CRP) at Week 12
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline to Week 12
Population: ITT analysis set participants with non-missing baseline and at least one post-baseline value were included; all observed data up to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 93 | 95 | 90 | 86 | 94
units on a scale | -1.08 [-1.35 to -0.82] | -1.59 [-1.85 to -1.33] | -2.09 [-2.37 to -1.82] | -2.51 [-2.78 to -2.23] | -1.71 [-1.96 to -1.45]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.007, Mixed Models Analysis; MMRM includes treatment, visit, treatment-by-visit interaction, stratification factors, and the baseline measurement as covariates; Least Squares (LS) Mean Difference = -0.51, 95% CI 2-sided [-0.87 to -0.14] — Response Rate Difference = ABBV-154 40mg - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Mixed Models Analysis; MMRM model includes treatment, visit, treatment-by-visit interaction, stratification factors, and the baseline measurement as covariates; Least Squares (LS) Mean Difference = -1.01, 95% CI 2-sided [-1.38 to -0.64] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -1.42, 95% CI 2-sided [-1.80 to -1.05] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -0.62, 95% CI 2-sided [-0.99 to -0.26] — Response Rate Difference = ABBV-154 340 E4W - Placebo

3. Secondary Outcome: Change in Clinical Disease Activity Index (CDAI) at Week 12
Description: CDAI is a composite index for assessing disease activity based on the sum of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and Physician's Global Assessment of Disease Activity (NRS). The total CDAI score ranges from 0 to 76 with higher scores indicating higher disease activity.
Time Frame: Baseline to Week 12
Population: Intent-to-treat analysis set participants with non-missing baseline and at least one post-baseline value were included; all observed data up to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 92 | 91 | 88 | 86 | 93
units on a scale | -14.21 [-16.81 to -11.60] | -18.77 [-21.41 to -16.13] | -22.21 [-24.94 to -19.48] | -25.62 [-28.31 to -22.93] | -19.50 [-22.06 to -16.94]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.014, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -4.56, 95% CI 2-sided [-8.21 to -0.92] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -8.01, 95% CI 2-sided [-11.70 to -4.31] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -11.41, 95% CI 2-sided [-15.10 to -7.73] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p = 0.004, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -5.29, 95% CI 2-sided [-8.89 to -1.69] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician's Global Assessment of Disease Activity (NRS)
     * Patient's Global Assessment of Disease Activity (NRS)
     * Patient's Assessment of Pain (NRS)
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
percentage of participants | 28.1 [19.1 to 37.1] | 52.7 [42.7 to 62.7] | 59.3 [49.3 to 69.2] | 74.4 [65.4 to 83.5] | 54.3 [44.2 to 64.3]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 24.7, 95% CI 2-sided [12.1 to 37.3] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 30.2, 95% CI 2-sided [17.4 to 42.9] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 45.4, 95% CI 2-sided [33.5 to 57.4] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 24.6, 95% CI 2-sided [11.9 to 37.3] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician's Global Assessment of Disease Activity (NRS)
     * Patient's Global Assessment of Disease Activity (NRS)
     * Patient's Assessment of Pain (NRS)
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
percentage of participants | 3.1 [0.0 to 6.6] | 9.2 [3.5 to 14.9] | 12.8 [6.1 to 19.6] | 13.3 [6.3 to 20.4] | 4.3 [0.2 to 8.3]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.031, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 6.5, 95% CI 2-sided [0.6 to 12.4] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 9.8, 95% CI 2-sided [2.7 to 17.0] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 10.9, 95% CI 2-sided [3.6 to 18.2] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p = 0.709, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 0.9, 95% CI 2-sided [-4.0 to 5.9] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

6. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Defined by DAS28 (CRP) <= 3.2 at Week 12
Description: Low disease activity (LDA) was defined as a DAS28 score less than or equal to 3.2. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS) and Physician's Global Assessment of Disease Activity (NRS), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
percentage of participants | 20.8 [12.7 to 29.0] | 38.9 [29.2 to 48.6] | 48.2 [38.0 to 58.3] | 53.3 [43.0 to 63.6] | 45.7 [35.7 to 55.8]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 16.9, 95% CI 2-sided [4.9 to 28.9] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 25.8, 95% CI 2-sided [13.5 to 38.1] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 31.5, 95% CI 2-sided [18.9 to 44.2] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 23.2, 95% CI 2-sided [11.0 to 35.4] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

7. Secondary Outcome: Percentage of Participants Achieving LDA Defined by CDAI <= 10 at Week 12
Description: Low disease activity based on CDAI is defined as a CDAI score less than or equal to 10. CDAI is a composite index for assessing disease activity based on the sum of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and Physician's Global Assessment of Disease Activity (NRS). The total CDAI score ranges from 0 to 76 with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
percentage of participants | 21.9 [13.6 to 30.1] | 36.8 [27.3 to 46.4] | 46.1 [36.0 to 56.2] | 46.7 [36.4 to 57.0] | 36.2 [26.5 to 45.9]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 14.1, 95% CI 2-sided [2.0 to 26.2] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 22.8, 95% CI 2-sided [10.0 to 35.5] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 24.3, 95% CI 2-sided [11.6 to 37.0] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p = 0.042, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 12.6, 95% CI 2-sided [0.5 to 24.7] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

8. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Defined by DAS28 (CRP) < 2.6 at Week 12
Description: Clinical remission was defined as a DAS28 (CRP) score less than 2.6. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
percentage of participants | 12.5 [5.9 to 19.1] | 18.4 [10.7 to 26.1] | 33.0 [23.5 to 42.6] | 37.8 [27.8 to 47.8] | 27.7 [18.6 to 36.7]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.296, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 5.1, 95% CI 2-sided [-4.4 to 14.6] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 19.5, 95% CI 2-sided [8.7 to 30.2] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 25.5, 95% CI 2-sided [14.3 to 36.7] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 14.1, 95% CI 2-sided [3.8 to 24.5] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

9. Secondary Outcome: Percentage of Participants Achieving CR Defined by CDAI <= 2.8 at Week 12
Description: Clinical Remission was defined by CDAI as a score less than or equal to 2.8. CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and Physician's Global Assessment of Disease Activity (NRS). The total CDAI score ranges from 0 to 76 with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 96 | 98 | 94 | 90 | 94
percentage of participants | 2.1 [0.0 to 4.9] | 9.2 [3.5 to 14.9] | 4.3 [0.2 to 8.3] | 4.4 [0.2 to 8.7] | 3.2 [0.0 to 6.7]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 7.1, 95% CI 2-sided [1.3 to 13.0] — Response Rate Difference = ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p = 0.424, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 2.0, 95% CI 2-sided [-2.8 to 6.8] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p = 0.303, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 2.6, 95% CI 2-sided [-2.3 to 7.5] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p = 0.551, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the stratification factors; Response Rate Difference = 1.3, 95% CI 2-sided [-2.9 to 5.4] — Response Rate Difference = ABBV-154 340 E4W - Placebo

10. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) to Week 12
Description: The Health Assessment Questionnaire - Disability Index is a participant-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W
Number analyzed (Participants) | 94 | 95 | 90 | 86 | 94
units on a scale | -0.08 [-0.19 to 0.03] | -0.26 [-0.36 to -0.15] | -0.33 [-0.45 to -0.22] | -0.41 [-0.52 to -0.29] | -0.29 [-0.39 to -0.18]
Statistical Analysis 1: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW; Test type: Superiority; p = 0.022, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -0.18, 95% CI 2-sided [-0.33 to -0.03] — ABBV-154 40mg EOW - Placebo
Statistical Analysis 2: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW; Test type: Superiority; p = 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -0.25, 95% CI 2-sided [-0.41 to -0.10] — Response Rate Difference = ABBV-154 150mg EOW - Placebo
Statistical Analysis 3: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -0.32, 95% CI 2-sided [-0.48 to -0.17] — Response Rate Difference = ABBV-154 340mg EOW - Placebo
Statistical Analysis 4: Comparison: Period 1 (Placebo-Controlled Period) Placebo vs Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W; Test type: Superiority; p = 0.007, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Least Squares (LS) Mean Difference = -0.21, 95% CI 2-sided [-0.36 to -0.06] — Response Rate Difference = ABBV-154 340mg E4W - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to end of study. Median time participants were followed was 85 days for all groups in Period 1. For each LTE group, the median time participants were followed was 412 days (Placebo-ABBV-154 150 mg EOW); 389 days (Placebo-ABBV-154 340 mg EOW); 390 days (ABBV-154 40 mg EOW); 402.5 days (ABBV-154 150 mg EOW), 404 days (ABBV-154 340 mg EOW), and 380 days (ABBV-154 340 mg E4W), respectively.
Description: All Randomized Population (N=473)
Groups:
- Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW: Participants in this group received placebo SC EOW for 12 weeks in the placebo-controlled period and then received ABBV-154 150mg SC EOW for 66 weeks in the LTE period.
- Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW: Participants in this group received placebo SC EOW for 12 weeks in the placebo-controlled period and then received ABBV-154 340mg SC EOW for 66 weeks in the LTE period.
Arm/Group | Period 1 (Placebo-Controlled Period) Placebo | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W | Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW | Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW | Period 2 (Extension Period) ABBV-154 40 mg EOW | Period 2 (Extension Period) ABBV-154 150 mg EOW | Period 2 (Extension Period) ABBV-154 340 mg EOW | Period 2 (Extension Period) ABBV-154 340 mg E4W
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/98 | 0/95 | 0/90 | 0/94 | 0/45 | 0/46 | 1/91 | 0/86 | 0/84 | 3/89
Serious Adverse Events (participants affected / at risk) | 2/96 | 4/98 | 6/95 | 5/90 | 3/94 | 3/45 | 6/46 | 7/91 | 8/86 | 10/84 | 9/89
Other Adverse Events (participants affected / at risk) | 25/96 | 43/98 | 26/95 | 26/90 | 27/94 | 31/45 | 25/46 | 54/91 | 56/86 | 52/84 | 47/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 (Placebo-Controlled Period) Placebo (N=96) | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW (N=98) | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW (N=95) | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW (N=90) | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W (N=94) | Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW (N=45) | Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW (N=46) | Period 2 (Extension Period) ABBV-154 40 mg EOW (N=91) | Period 2 (Extension Period) ABBV-154 150 mg EOW (N=86) | Period 2 (Extension Period) ABBV-154 340 mg EOW (N=84) | Period 2 (Extension Period) ABBV-154 340 mg E4W (N=89)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROLOGICAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPPORTUNISTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Q FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STROKE IN EVOLUTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 (Placebo-Controlled Period) Placebo (N=96) | Period 1 (Placebo-Controlled Period) ABBV-154 40 mg EOW (N=98) | Period 1 (Placebo-Controlled Period) ABBV-154 150 mg EOW (N=95) | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg EOW (N=90) | Period 1 (Placebo-Controlled Period) ABBV-154 340 mg E4W (N=94) | Period 2 (Extension Period) Placebo to ABBV-154 150mg EOW (N=45) | Period 2 (Extension Period) Placebo to ABBV-154 340mg EOW (N=46) | Period 2 (Extension Period) ABBV-154 40 mg EOW (N=91) | Period 2 (Extension Period) ABBV-154 150 mg EOW (N=86) | Period 2 (Extension Period) ABBV-154 340 mg EOW (N=84) | Period 2 (Extension Period) ABBV-154 340 mg E4W (N=89)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (5) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 5 (6) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 5 (7) | 1 (1) | 2 (2)
INJECTION SITE BRUISING (General disorders) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (13) | 2 (3) | 2 (4) | 2 (2) | 6 (6)
INJECTION SITE DISCOLOURATION (General disorders) | 0 (0) | 3 (4) | 1 (2) | 4 (4) | 1 (1) | 4 (5) | 3 (5) | 2 (2) | 5 (5) | 3 (3) | 3 (3)
INJECTION SITE ERYTHEMA (General disorders) | 1 (3) | 3 (7) | 1 (1) | 3 (6) | 6 (7) | 2 (3) | 3 (9) | 7 (35) | 3 (14) | 5 (8) | 5 (8)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 6 (6) | 3 (3) | 3 (3) | 0 (0)
BRONCHITIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 2 (2) | 2 (2) | 6 (6)
COVID-19 (Infections and infestations) | 1 (1) | 13 (13) | 5 (5) | 2 (2) | 7 (7) | 12 (12) | 8 (8) | 15 (17) | 15 (16) | 17 (18) | 16 (17)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 4 (6)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 2 (2) | 4 (5) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 9 (11) | 11 (13) | 6 (6) | 11 (15)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 3 (3) | 3 (3) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 4 (4) | 9 (11) | 5 (5) | 6 (6) | 8 (10) | 12 (13) | 7 (7)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 8 (10) | 5 (10) | 3 (3) | 6 (8) | 8 (10) | 5 (5)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 3 (3) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 3 (3) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 8 (8) | 3 (3) | 2 (2)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (6) | 2 (2) | 1 (1) | 2 (2) | 5 (6) | 4 (6) | 10 (12) | 11 (14) | 5 (5) | 8 (10)
HEADACHE (Nervous system disorders) | 3 (3) | 4 (4) | 3 (3) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 5 (5) | 3 (5) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (5) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 4 (4) | 4 (9) | 3 (3) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04888585/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT04888585/SAP_001.pdf